CLINICAL TRIAL: NCT04343521
Title: Quantifying the Epidemiological Impact of Targeted Indoor Residual Spraying on Aedes-borne Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Gonzalo Vazquez-Prokopec, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00108666; 1U01AI148069-01 (NIH)
Record Dates: First submitted 2020-04-09; First posted 2020-04-13 (Actual); Results first posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: Aedes-borne Diseases; Dengue; Chikungunya; Zika
Keywords: Targeted Indoor Residual Spraying; Children; Dengue virus (DENV); Chikungunya virus (CHIKV); Zika virus (ZIKV); Ae. aegypti mosquito
MeSH Terms: conditions — Mosquito-Borne Diseases; Dengue; Chikungunya Fever; Zika Virus Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted Indoor Residual Spraying (TIRS) (Experimental): All households in Targeted Indoor Residual Spraying (TIRS) clusters will be offered the intervention, and children in households that consent to TIRS will be recruited into this study arm.
  Interventions: Other: Targeted Indoor Residual Spraying (TIRS)
- Routine Aedes-borne Virus (ABV) Prevention and Control (No Intervention): Households in the control clusters receive routine Aedes-borne virus (ABV) prevention and control, without Targeted Indoor Residual Spraying (TIRS). Children in the control households will be recruited into this study arm.

INTERVENTIONS:
Other: Targeted Indoor Residual Spraying (TIRS) — Spraying of insecticide Actellic 300CS will start in May or June extending for 1 to 2 months. Residents will be asked to temporarily leave the house during treatment and wait half an hour to one hour for the product to dry before re-entering the house. Insecticide application will follow strict protocol developed by the Centers for Disease Control and Prevention (CDC), Emory University, and the Universidad Autónoma de Yucatán.
  Other Names: Actellic 300CS
  Arms: Targeted Indoor Residual Spraying (TIRS)

SUMMARY:
The objective of this trial is evaluate the efficacy of Targeted Indoor Residual Spraying (TIRS) in preventing symptomatic disease caused by Aedes-borne diseases (ABDs) in children 2 to 15 years of age in the city of Merida, Yucatan State, Mexico.

DETAILED DESCRIPTION:
Contemporaneous urban vector control (truck-mounted ultra-low volume spraying, thermal fogging, larviciding) has failed to contain dengue epidemics and to prevent the global range expansion of Aedes-borne diseases (ABDs: dengue, chikungunya, zika). Part of the challenge in sustaining effective ABD control emerges from the remarkable paucity of evidence about the epidemiological impact of any vector control method. Furthermore, the classic deployment of interventions in response to clinical cases fails to account for the important contribution of out-of-home human mobility and asymptomatic infections.

The trial will be conducted in the city of Merida extending ongoing longitudinal cohort to follow a population of 4,600 children 2-15 years old randomly allocated to receive either TIRS treatment or not. If efficacious, TIRS will drive a paradigm shift in Aedes control by: considering Ae. aegypti behavior to rationally guide insecticide applications; the change to preventive control (pre- ABD transmission season rather than in response to symptomatic cases); the use of third generation insecticides to which Ae. Aegypti is susceptible.

ELIGIBILITY:
Inclusion Criteria:

Household Level Inclusion Criteria:

* Household is located within the bounds of a study cluster (5x5 city-block clusters)
* City block has at least 60% premises that are residential

Individual Level Inclusion Criteria:

* 2 or more and up to 15 years of age at the time of initial enrollment
* Living in a house that consented to TIRS (for children in TIRS cluster)

Exclusion Criteria:

Household Level Exclusion Criteria:

* Households where study personnel identify a security risk (i.e., site where drugs are sold, residents are always drunk or hostile)
* Sites where no residents spend time during the day (i.e. work 7days a week outside the home)
* Inability for a resident to provide informed consent
* Non-residential places (e.g., businesses, schools, markets, etc.)

Individual Level Exclusion Criteria:

* Less than 2 years of age or more than 15 years of age at the time of enrollment
* Not living in a house that consented to TIRS (for children in TIRS cluster)
* Having a medical condition that prevents implementation of study procedures
* Temporary visitor to household
* Plans to leave study area within next 12 months

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4461 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2024-04-28 (Actual); Study Completion 2024-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Vazquez Prokopec, MD, Principal Investigator — Emory University
Locations (1):
- Universidad Autonoma de Yucatan, Mérida, Yucatán, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data that underlie the results reported in publications of this study will be available for sharing with other researchers.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available for sharing starting one year following conclusion of the trial, with no end date.
Access Criteria: Investigators wanting to share data from this study should provide a methodologically sound proposal. Data will be shared with other researchers in order for them to achieve aims in the approved proposal. Proposals should be directed to lwaller@emory.edu. To gain access, data requesters will need to sign a data access agreement.

REFERENCES:
- [Background] Manrique-Saide P, Dean NE, Halloran ME, Longini IM, Collins MH, Waller LA, Gomez-Dantes H, Lenhart A, Hladish TJ, Che-Mendoza A, Kirstein OD, Romer Y, Correa-Morales F, Palacio-Vargas J, Mendez-Vales R, Perez PG, Pavia-Ruz N, Ayora-Talavera G, Vazquez-Prokopec GM. The TIRS trial: protocol for a cluster randomized controlled trial assessing the efficacy of preventive targeted indoor residual spraying to reduce Aedes-borne viral illnesses in Merida, Mexico. Trials. 2020 Oct 8;21(1):839. doi: 10.1186/s13063-020-04780-7. PMID 33032661
- [Background] Che-Mendoza A, Gonzalez-Olvera G, Medina-Barreiro A, Arisqueta-Chable C, Bibiano-Marin W, Correa-Morales F, Kirstein OD, Manrique-Saide P, Vazquez-Prokopec GM. Efficacy of targeted indoor residual spraying with the pyrrole insecticide chlorfenapyr against pyrethroid-resistant Aedes aegypti. PLoS Negl Trop Dis. 2021 Oct 4;15(10):e0009822. doi: 10.1371/journal.pntd.0009822. eCollection 2021 Oct. PMID 34606519
- [Background] Dzul-Manzanilla F, Correa-Morales F, Che-Mendoza A, Palacio-Vargas J, Sanchez-Tejeda G, Gonzalez-Roldan JF, Lopez-Gatell H, Flores-Suarez AE, Gomez-Dantes H, Coelho GE, da Silva Bezerra HS, Pavia-Ruz N, Lenhart A, Manrique-Saide P, Vazquez-Prokopec GM. Identifying urban hotspots of dengue, chikungunya, and Zika transmission in Mexico to support risk stratification efforts: a spatial analysis. Lancet Planet Health. 2021 May;5(5):e277-e285. doi: 10.1016/S2542-5196(21)00030-9. PMID 33964237
- [Background] Kirstein OD, Ayora-Talavera G, Koyoc-Cardena E, Chan Espinoza D, Che-Mendoza A, Cohuo-Rodriguez A, Granja-Perez P, Puerta-Guardo H, Pavia-Ruz N, Dunbar MW, Manrique-Saide P, Vazquez-Prokopec GM. Natural arbovirus infection rate and detectability of indoor female Aedes aegypti from Merida, Yucatan, Mexico. PLoS Negl Trop Dis. 2021 Jan 4;15(1):e0008972. doi: 10.1371/journal.pntd.0008972. eCollection 2021 Jan. PMID 33395435
- [Background] Dzib-Florez S, Ponce-Garcia G, Medina-Barreiro A, Gonzalez-Olvera G, Contreras-Perera Y, Del Castillo-Centeno F, Ahmed AMM, Che-Mendoza A, McCall PJ, Vazquez-Prokopec G, Manrique-Saide P. Evaluating Over-the-Counter Household Insecticide Aerosols for Rapid Vector Control of Pyrethroid-Resistant Aedes aegypti. Am J Trop Med Hyg. 2020 Nov;103(5):2108-2112. doi: 10.4269/ajtmh.20-0515. PMID 32748782
- [Derived] Dean NE, Crisp AM, Che-Mendoza A, Kirstein OD, Barrera-Fuentes GA, Earnest JT, Puerta-Guardo HN, Collins MH, Pavia-Ruz N, Ayora-Talavera G, Gonzalez-Olvera G, Medina-Barreiro A, Bibiano-Marin W, Jabbarzadeh S, Halloran ME, Longini IM Jr, Lenhart A, Waller LA, Correa-Morales F, Palacio-Vargas J, Gomez-Dantes H, Manrique-Saide P, Vazquez-Prokopec GM. Randomized Trial of Targeted Indoor Spraying to Prevent Aedes-Borne Diseases. N Engl J Med. 2025 Oct 9;393(14):1387-1398. doi: 10.1056/NEJMoa2501069. PMID 41061233
- See also: link to project website — https://www.prokopeclab.org/tirs-1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants are children from households in the study clusters in Merida, Yucatan, Mexico. Participant enrollment began November 3, 2020 and all follow-up assessments were completed by April 28, 2024.
Units Other Than Participants: Households
Groups:
- Targeted Indoor Residual Spraying (TIRS): Children residing in households located in Targeted Indoor Residual Spraying (TIRS) clusters that were offered the intervention.
  During Targeted Indoor Residual Spraying (TIRS), spraying of the insecticide Actellic 300CS began in May or June extending for 1 to 2 months. Residents were asked to temporarily leave the house during treatment and wait half an hour to one hour for the product to dry before re-entering the house. Insecticide application followed a strict protocol developed by the Centers for Disease Control and Prevention (CDC), Emory University, and the Universidad Autónoma de Yucatán.
- Routine Aedes-borne Virus (ABV) Prevention and Control: Children residing in households located in routine Aedes-borne virus (ABV) prevention and control clusters, without Targeted Indoor Residual Spraying (TIRS).
Period: Overall Study
Arm/Group | Targeted Indoor Residual Spraying (TIRS) | Routine Aedes-borne Virus (ABV) Prevention and Control
Started | 2239; 13487 Households | 2222; 13486 Households
Completed | 1835; 10472 Households | 1718; 13486 Households
Not Completed | 404; 3015 Households | 504; 0 Households
Not completed — Adverse Event | 0 | 2
Not completed — Death | 1 | 2
Not completed — Lost to follow-up due to moving from the cluster | 327 | 393
Not completed — Withdrawal by Subject | 70 | 95
Not completed — Withdrawal by study team | 6 | 12

BASELINE CHARACTERISTICS:
Groups:
- Targeted Indoor Residual Spraying (TIRS): Children residing in households located in Targeted Indoor Residual Spraying (TIRS) clusters that were offered the intervention.
- Total: Total of all reporting groups
Arm/Group | Targeted Indoor Residual Spraying (TIRS) | Routine Aedes-borne Virus (ABV) Prevention and Control | Total
Number analyzed (Participants) | 2239 | 2222 | 4461
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2239 | 2222 | 4461
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1108 | 1053 | 2161
  Male | 1131 | 1169 | 2300
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2239 | 2222 | 4461
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Mexico | 2239 | 2222 | 4461

OUTCOME MEASURES:

1. Primary Outcome: Number of Symptomatic Participants Testing Positive for Aedes-borne Virus Infections That Are Laboratory Confirmed or Serologically
Description: The number of symptomatic children with laboratory confirmed, by reverse transcription-polymerase chain reaction (RT-PCR) or immunoglobulin M/ immunoglobulin G (IgM/IgG) enzyme-linked immunosorbent assay (ELISA), Aedes-borne Viruses infections. The number of any Aedes-borne virus infection during three seasons of high transmission is described, as well as the number of Dengue virus (DENV), Chikungunya virus (CHIKV), Zika virus (ZIKV) and coinfections.
Time Frame: 18 months of active surveillance during high transmission seasons (each 6 months in duration) during 3 years (July through December in 2021, 2022, and 2023)
Population: This analysis includes symptomatic children who were tested for Andes-borne viruses during high transmission seasons.
Measure: Count of Participants; unit: Participants
Arm/Group | Targeted Indoor Residual Spraying (TIRS) | Routine Aedes-borne Virus (ABV) Prevention and Control
Number analyzed (Participants) | 402 | 423
Participants
  Number of Children Testing Positive for All Aedes-borne Viruses | 213 | 209
  Number of Children Testing Positive for DENV | 151 | 146
  Number of Children Testing Positive for CHIKV | 1 | 0
  Number of Children Testing Positive for ZIKV | 39 | 55
  Number of Children Testing Positive for Coinfection | 22 | 8

2. Secondary Outcome: Number Positive Tests of Laboratory Confirmed Aedes-borne Viruses Infections By Season
Description: Number of laboratory confirmed (IgG ELISA and neutralization testing) Aedes-borne Viruses (DENV, CHIKV and ZIKV) in annual surveillance samples.
Time Frame: Up to 36 months, during serosurvey seasons 2021-2022, 2022-2023, and 2023-2024
Population: The population analyzed includes children living in study households where annual surveillance sampling for Aedes-borne viruses occurred.
Measure: Count of Units; unit: Number of Tests
Units Other Than Participants: Number of Tests
Arm/Group | Targeted Indoor Residual Spraying (TIRS) | Routine Aedes-borne Virus (ABV) Prevention and Control
Number analyzed (Participants) | 2239 | 2222
Number analyzed (Number of Tests) | 1933 | 1932
Number of Tests
  Number of Positive Tests for all Aedes-borne Viruses During 2021-2022 Season: number analyzed (Participants) | 1933 | 1932
  Number of Positive Tests for all Aedes-borne Viruses During 2021-2022 Season: number analyzed (Number of Tests) | 589 | 591
  Number of Positive Tests for all Aedes-borne Viruses During 2021-2022 Season | 36 | 39
  Number of Positive Tests for all Aedes-borne Viruses During 2022-2023 Season: number analyzed (Participants) | 1351 | 1415
  Number of Positive Tests for all Aedes-borne Viruses During 2022-2023 Season: number analyzed (Number of Tests) | 683 | 683
  Number of Positive Tests for all Aedes-borne Viruses During 2022-2023 Season | 216 | 166
  Number of Positive Tests for all Aedes-borne Viruses During 2023-2024 Season: number analyzed (Participants) | 1116 | 1127
  Number of Positive Tests for all Aedes-borne Viruses During 2023-2024 Season: number analyzed (Number of Tests) | 661 | 658
  Number of Positive Tests for all Aedes-borne Viruses During 2023-2024 Season | 169 | 204

3. Secondary Outcome: Ae. Aegypti Mosquito Infection Rate With Aedes-borne Viruses (DENV, CHIKV and ZIKV)
Description: Ae. aegypti mosquito infection rate with Aedes-borne Viruses (DENV, CHIKV and ZIKV) assessed by the number of positive RT-PCR tests. Infection is mosquitoes is analyzed by collecting binary data (a mosquito pool is either infected or not) and transforming that into minimum infection rates (MIR) with the calculation: (1/number of mosquitoes in the pool) times 1000. Households were randomly selected for testing; houses were eligible for testing if they were located within the central blocks and had at least one child enrolled in the study.
Time Frame: Up to 6 months (mosquito pools were collected during the 6 months post TIRS spraying samplings in 2021)
Population: This analysis includes households where mosquito sampling occurred. Individual participants were not analyzed. Only households contributed data.
Measure: Count of Units; unit: Households samples
Units Other Than Participants: Households samples
Groups:
- Households in Targeted Indoor Residual Spraying (TIRS) Clusters: Households located in Targeted Indoor Residual Spraying (TIRS) clusters that were offered the intervention.
- Households in Routine Aedes-borne Virus (ABV) Prevention and Control Clusters: Households located in routine Aedes-borne virus (ABV) prevention and control clusters, without Targeted Indoor Residual Spraying (TIRS).
Arm/Group | Households in Targeted Indoor Residual Spraying (TIRS) Clusters | Households in Routine Aedes-borne Virus (ABV) Prevention and Control Clusters
Number analyzed (Participants) | NA | NA
Number analyzed (Households samples) | 160 | 160
Households samples | 0 | 0

4. Secondary Outcome: Ae. Aegypti Indoor Entomological Index of Adult Mosquito Abundance
Description: The Ae. aegypti indoor entomological index of adult mosquito presence/abundance is calculated as the number of adult mosquitoes per house. Higher values mean that more mosquitoes are found within houses.
Time Frame: Up to 36 months starting at the first TIRS application
Measure: Mean (Standard Deviation); unit: mosquitoes/house
Units Other Than Participants: Households
Arm/Group | Targeted Indoor Residual Spraying (TIRS) | Routine Aedes-borne Virus (ABV) Prevention and Control
Number analyzed (Participants) | 2239 | 2222
Number analyzed (Households) | 13487 | 13486
mosquitoes/house | 0.61 (1.1) | 1.39 (2.1)

5. Secondary Outcome: Ae. Aegypti Indoor Entomological Index of Female Mosquito Abundance
Description: The Ae. aegypti indoor entomological index of female mosquito presence/abundance is calculated as the number of female mosquitoes per house. Higher values mean that more mosquitoes are found within houses.
Time Frame: Up to 36 months starting at first TIRS application
Measure: Mean (Standard Deviation); unit: mosquitoes/house
Units Other Than Participants: Households
Arm/Group | Targeted Indoor Residual Spraying (TIRS) | Routine Aedes-borne Virus (ABV) Prevention and Control
Number analyzed (Participants) | 2239 | 2222
Number analyzed (Households) | 13487 | 13486
mosquitoes/house | 0.29 (0.9) | 0.65 (1.9)

6. Secondary Outcome: Ae. Aegypti Indoor Entomological Index of Bloodfed Female Mosquito Abundance
Description: The Ae. aegypti indoor entomological index of bloodfed female mosquito presence/abundance is calculated as the number of bloodfed female mosquitoes per house. Higher values mean that more mosquitoes are found within houses.
Time Frame: Up to 36 months starting at first TIRS application
Measure: Mean (Standard Deviation); unit: mosquitoes/house
Units Other Than Participants: Households
Arm/Group | Targeted Indoor Residual Spraying (TIRS) | Routine Aedes-borne Virus (ABV) Prevention and Control
Number analyzed (Participants) | 2239 | 2222
Number analyzed (Households) | 13487 | 13486
mosquitoes/house | 0.25 (0.92) | 0.53 (0.94)

7. Secondary Outcome: Number of Households Where the Head of Household Would Recommend the Intervention
Description: Acceptability of the intervention is determined through household surveys, for households that received the intervention. Acceptability is assessed as the number of households where the head of that household would recommend the intervention to others.
Time Frame: Post-intervention (up to 41 months and 26 days after the start of the intervention)
Population: This analysis includes households in TIRS clusters where the head of the household completed the household survey.
Measure: Count of Units; unit: Households
Units Other Than Participants: Households
Groups:
- Households With Targeted Indoor Residual Spraying (TIRS): Households located in Targeted Indoor Residual Spraying (TIRS) clusters that were offered the intervention.
Arm/Group | Households With Targeted Indoor Residual Spraying (TIRS)
Number analyzed (Participants) | NA
Number analyzed (Households) | 2250
Households | 2160

8. Secondary Outcome: Number of Households With a Resident That Had a Reaction to the Insecticide
Description: Safety of the intervention is assessed as the number of households receiving the TIRS intervention that had evidence of a household resident having a reaction possibly related to the insecticide, which was assessed and confirmed by study doctors.
Time Frame: Post-intervention (up to 41 months and 26 days after the start of the intervention)
Population: This analysis includes households in TIRS clusters where the head of the household completed the household survey.
Measure: Count of Units; unit: Households
Units Other Than Participants: Households
Arm/Group | Households With Targeted Indoor Residual Spraying (TIRS)
Number analyzed (Participants) | NA
Number analyzed (Households) | 2250
Households | 2

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the time when individuals gave consent to participate in the study and continued through the final assessment (up to 41 months and 26 days).
Arm/Group | Targeted Indoor Residual Spraying (TIRS) | Routine Aedes-borne Virus (ABV) Prevention and Control
All-Cause Mortality (participants affected / at risk) | 1/2239 | 2/2222
Serious Adverse Events (participants affected / at risk) | 0/2239 | 2/2222
Other Adverse Events (participants affected / at risk) | 6/2239 | 4/2222
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Targeted Indoor Residual Spraying (TIRS) (N=2239) | Routine Aedes-borne Virus (ABV) Prevention and Control (N=2222)
Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Aplastic anemia secondary to parvovirus and rickettsiosis infection (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Targeted Indoor Residual Spraying (TIRS) (N=2239) | Routine Aedes-borne Virus (ABV) Prevention and Control (N=2222)
Admission to emergency room due to dengue with warning signs (Infections and infestations) | 3 | 2
Admission to emergency room due to suspected dengue with warning signs (Infections and infestations) | 1 | 2
Mild allergic reaction (General disorders) | 1 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT04343521/Prot_SAP_001.pdf
  • Informed Consent Form (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/21/NCT04343521/ICF_000.pdf